CLINICAL TRIAL: NCT04464538
Title: Sedentary Behaviour and Cognitive Function in Community Dwelling Older People: A Feasibility Study
Brief Title: Reducing Sedentary Behaviour and Cognition in Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Collaborators: Cambridgeshire and Peterborough NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Olawale Olanrewaju, Principal Investigator, Anglia Ruskin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRAS280073
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Mild Cognitive Impairment
Keywords: Sedentary behaviour; Cognitive function; Feasibility study; Older adults
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Unblinded, single-centre randomized feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health information (Placebo Comparator): Participants in the control group will complete baseline measures, and then they will receive written information on the benefits of increasing activity levels. This advice will be given in accordance with NHS guide on physical health.
  Interventions: Other: Information leaflet
- Group education session and individualised coaching (online) (Experimental): Participants assigned to the WALC-R intervention will attend a virtual baseline educational group session which will include a maximum of five people. The aim of the sessions will be to introduce the basics of the benefits of walking for exercise and why exercise is beneficial, as well as to give information, support and motivation to help participants to independently walk more in their daily routines.The group session will also include goal setting, in which participants will be encouraged to set their own daily walking targets to increase their habitual levels of walking. All participants will be given a pedometer to self-monitor how far they walk and a diary to record activity context throughout the intervention daily. Participants will meet briefly (20-30 minutes) via the internet with an assigned coach every 2 weeks.
  Interventions: Behavioral: WALC-R

INTERVENTIONS:
Behavioral: WALC-R — Initial group education session and individualized coaching (remote)
  Arms: Group education session and individualised coaching (online)
Other: Information leaflet — Participants in the control group will complete baseline measures, and then they will receive written information on the benefits of increasing activity levels. This advice will be given in accordance with NHS guide on physical health.
  Arms: Health information

SUMMARY:
Introduction Sedentary behaviour refers to activities of low energy expenditure in lying and sitting positions. Examples include driving, watching television, playing cards, puzzles and working on a computer. Studies suggest that between 60% of older people world-wide reported sitting for more than four hours per day. Sedentary behaviour increases as older people become older, have problems with cognition and when they are very ill. Excessive participating in sedentary behaviours is associated with an increased risk of heart problem, cancer death and diabetes. However, we do not know for certain whether or not participating in sedentary behaviour could cause poorer cognition.

What does the study hope to achieve?

This feasibility study will test whether the main study, which is planned for later, is workable with regards to the following:

* Will reducing sedentary behaviour using our online health coaching intervention (WALC-R) be acceptable to research participants and caregivers?
* How many participants can be successfully recruited to the future trial?
* What is the rate of adverse event associated with proposed study intervention?

Method:

This is a 13-week randomised feasibility study. We will randomly assign study participants to either the health coaching intervention (WALC-R) or receiving health guidelines on recommended physical activity. We aim to recruit 40 participants aged 50 and over who have been diagnosed with Mild Cognitive Impairment.

The future main study will be larger and test whether:

• 'WALC-R', an online intervention designed to reduce participation in sedentary behaviour can improve cognitive function in older people with Mild Cognitive Impairment compared with providing an information sheet about physical activity.

DETAILED DESCRIPTION:
Background / Rationale The participation in sedentary behaviors is high among the older population and increases with age co-morbidities and cognitive decline. 60% of older adults world-wide reported sitting for more than four hours per day and when device-measured, 67% of the older population were sedentary for more than 8.5 hours in their waking day (Harvey et al., 2015). Further, recent policies of confinement and restriction stipulated by various governments in response to the global COVID-19 pandemic is likely to encourage greater participation in sedentary behavior (Ricci et al., 2020). There is evidence of deleterious health implications of sedentary behaviors, with possible independent associations with all-cause mortality, cardiovascular disease mortality, cardiovascular disease incidence, cancer mortality, and type 2 diabetes incidence(Biswas and Alter, 2015). However, the associations between sedentary behaviors and cognitive health are less clear and inconclusive. A recent systematic review of 18 studies found inconclusive evidence on the overall and independent associations between sedentary behaviors and cognitive function in older adults (Olanrewaju et al., 2020). The review highlighted the lack of quality and intervention studies of effect as one of the limitations of existing evidence.

There is some evidence that non-exercise and physical activity interventions could be effective in reducing sedentary behaviors in older adults. A review of strategies to reduce sedentary behavioural among adults found that the most promising interventions used behavioural change techniques such as self-monitoring and problem solving(Gardner et al., 2016). A recent meta-analysis of digital behavior change interventions (DBCI) in older adults suggested that using platforms such as mobile applications, websites, wearable devices reduced sedentary time by 58 minutes per day (SMD = -0.45; 95%CI -0.69, -0.19; p < 0.001) (Stockwell et al., 2019). A separate systematic review of interventions to reduce sedentary behavior in non-working older adults found that interventions which incorporated goal setting, individualized feedback, motivational sessions reduced objectively measured sitting time by 3.2%-5.3% of waking time or up to 54 minutes per day (Aunger et al., 2018).

The WALC intervention (Walk; Address sensations; Learn; Cue) was originally designed to motivate community-dwelling older adults to increase physical activity and is based on Social Cognitive theory (Resnick, 2001). The WALC intervention is not a walking/physical activity group, rather, a forum where the concept of sedentary behavior and strategies to reduce these behaviours are coached. The WALC intervention has been validated in several studies for use in the older population and people living with schizophrenia and more recently with serious mental illness (Beebe and Smith, 2010; Resnick et al., 2007; Williams et al., 2019). This study proposes to adopt the WALC intervention, which incorporates elements of the COM-B behavioral change model to address capability, opportunity, and motivational barriers to reduce sedentary behavior (Michie et al., 2011). Unlike original and previous versions of the WALC intervention, we propose to deliver our intervention (WALC-R) remotely via the internet. The WALC-R will consist of a group initial education session, fortnightly health coaching sessions, and self-monitoring of daily activity levels using pedometer and diary. There is no evidence on the effectiveness of non-exercise, sedentary behavior-reducing intervention on cognitive function in the older population. Therefore, we propose to test the feasibility of a remotely delivered health coaching intervention in older adults at risk of cognitive decline with a view to test for effectiveness on cognitive function in a later study.

Aim To test the feasibility, acceptability and costs of delivering a virtual health coaching intervention via the internet in community dwelling older people. This present proposal aims to pave the way for a future randomized controlled trial by resolving key uncertainties in its planning. The purpose of the future trial will be to test whether WALC-R intervention compared with providing information about physical activity can improve cognitive function in older adults with Mild Cognitive Impairment.

Objectives

1. To determine the acceptability of intervention to participants
2. To determine feasibility of study with respect to the following:

   1. Number of eligible patients
   2. Recruitment and retention rates
   3. Adherence / compliance rates
   4. Collection of potential outcome measures for future trial (completion rates and time)
3. To determine the costs associated with delivering intervention
4. To determine rate of adverse events in both groups.

Methods- Randomized Feasibility Study

Study design This will be a 13 week unblinded, single-centre randomized feasibility study. The intervention is comprised of an initial group education session, fortnightly coaching sessions and the provision of a pedometer and diary to enable participants monitor their daily physical activity. Participants in the control group will receive information leaflets which outlines the benefit of being physically active. The design will adhere to the Consolidated Standards of Reporting Trials statement (CONSORT).

Setting and Participants The study will be conducted remotely in the community settings of service users from Cambridgeshire and Peterborough NHS Foundation Trust (CPFT). Prior to starting permissions will be sought from local Research Ethics Committees (REC), CPFT Research and Development team and the National Research Authority.

Sampling Strategy Eligible patients who attend the memory clinics and / or receive support from the older people mental health and healthy ageing services in Cambridgeshire and Peterborough NHS Foundation Trust will be invited to participate.

Recruitment / Screening Potential participants would be primarily sought from the community mental health, living well, memory services and general practitioners in Cambridgeshire and Peterborough. A member of the clinical team will screen for potential participants for initial eligibility (from medical notes, clinic records and/or clinical consultations) and, if appropriate, given information about the trial. The clinician will then arrange an appointment to discuss the trial, along with the opportunity to ask any questions. The researcher will give people 24 hours to decide if they would like to participate. If they are happy with the information they receive, they will be contacted by a member of the research team to give informed consent. This study proposes to recruit patients with mild cognitive impairment. Therefore a mental capacity test will be conducted during the process of consent to ensure that participants understand, retain and weigh up the information available to make a decision about consenting. Participants' general practitioners will be informed about their enrolment onto the study. Once enrolled, participants will be asked to wear an accelerometer for 7 days. Each participant will be reimbursed £10 for wearing the accelerometer. After completion of the baseline measures, the participants will be informed of their allocation status.

Proposed sample size and Justification Total sample sizes between 24 and 50 have been recommended for feasibility studies. (18-20). Based on these recommendations, the study proposes to enroll 40 participants, a target sample of 24 (12 per group) after factoring a 40% drop-out rate.

Randomization, Post-randomization withdrawals and exclusions This study proposes a simple randomization of participants into intervention and control arms. Randomization process will be overseen by the researcher using freely available software from Sealed Envelope: https://www.sealedenvelope.com/help/simple-randomiser/students/. Participants will be randomly allocated to receive either 'WALC-R' (intervention group) or information on recommended physical activity for older adults (control group). Approximately 5 participants will be randomized each month over 8 months. Subjects may discontinue participation in the trial intervention and/or the trial at any time. Unless a subject explicitly withdraws their consent, they will be followed-up wherever possible and data collected as per the protocol until the end of the trial. Documentation will be completed on withdrawal to confirm the date and reason for withdrawal.

Summary of Intervention Initial group education session (online) Participants assigned to the WALC-R intervention will attend a virtual baseline educational group session which will include a maximum of five people. The aim of the sessions will be to introduce the basics of the benefits of walking for exercise and why exercise is beneficial, as well as to give information, support and motivation to help participants to independently walk more in their daily routines. In the group sessions, we will also introduce the concept of sedentary behaviour and the harms and strategies to sit less and move more, including disrupting prolonged periods of sitting. At the educational session, researchers will have information on the participants' habitual levels of physical activity obtained from baseline data collection. The group session will also include goal setting, in which participants will be encouraged to set their own daily walking targets to increase their habitual levels of walking. All participants will be given a pedometer to self-monitor how far they walk and a diary to record activity context throughout the intervention daily.

Continuing support and coaching (online) Participants will meet briefly (20-30 minutes) via the internet with an assigned worker (i.e., their coach) every 2 weeks. The participant and coach will review the participant's walking calendar and address any barriers to and facilitators of engaging in physical activity and reducing sedentary behaviour.

Control condition Participants in the control group will complete baseline measures, and then they will receive written information on the benefits of increasing activity levels. This advice will be given in accordance with NHS guide on physical health.

Follow-up assessment The follow-up assessment will be undertaken at the end of the intervention after 13 weeks. At follow-up, all measures will be repeated (apart from sociodemographic information). Each participant will receive a £10 voucher for wearing an accelerometer. These assessments will be done by a research worker who is blind to allocation status.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling adults aged 50+ years.
* Doctor diagnosis of Mild Cognitive Impairment OR MCI diagnosis which meets Petersen Criteria.
* Participants must have a working knowledge of English.
* Participants must be able to provide informed consent.

Exclusion Criteria:

* Individuals diagnosed by doctor with dementia.
* Individuals diagnosed with severe mental health conditions and substance use disorders e.g. alcohol or drug abuse in within the last year.
* Individuals with diagnosed neurological conditions.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of intervention assessed by semi-structured interviews | Week 13
  Acceptability of study intervention will be qualitatively assessed at the end of week 13 via semi-structured interviews with study participants.
Recruitment rate | Week 13
  Proportion of target recruit sample achieved throughout study duration.
Completeness of intervention | Week 13
  Proportion of participants recruited into the study who completed the intervention.
Adverse event rate | Week 13
  Proportion of people recruited into the study who sustained adverse events.

SECONDARY OUTCOMES:
Device measured sedentary behaviour | Week 1 and 13
  Sedentary behaviour and physical activity time per day will be recorded using ActivPAL inclinometer.All participants will be required to wear the ActivPAL continuously for at least 7 days at baseline that will measure habitual sedentary behaviour and walking activity each day (Edwardson et al., 2017). The inclinometer will record how many minutes per day each participant is sedentary and engages in light, moderate and vigorous physical activities. A recording is made of each 60-second period (called an 'epoch'), and this is classified as being sedentary or light, moderate or vigorous physical activity. The researcher will collect data on the total minutes of sedentary behaviour per day, number of disruptions in sedentary behaviour and total time spent in physical activity (minutes per day in light, moderate and vigorous activity).
Self reported sedentary behaviour assessed using the Sedentary Behaviour Questionnaire | Week 1 and 13
  Participants will complete a survey questionnaire about weekly time spent participating in selected sedentary behaviours such as watching television and sitting (Rosenberg et al., 2010). The options for respondents include 'None', <=15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6+ hours.
Verbal fluency assessed using the Controlled and Oral Word Association Test (COWAT) | Week 1 and 13
  The researcher will test participant's verbal fluency (cognitive function) using the Controlled and Oral Word Association Test. The scores represent the number of correct words provided in 60 seconds. Higher scores represent better verbal fluency ability and vice versa.
Perceived quality of life using the EuroQol five-dimension questionnaire (EQ-5D) | Week 1 and 13
  The participants will self- rate their health using five dimensions provided (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and five response levels: no problems, slight, moderate, severe, unable to/extreme problems. The EQ- Visual Analogue Scale(VAS) records the respondent's overall current health (0-100). Higher VAS scores represent best perceived health and vice versa.
Pre-morbid intelligence | Week 1 and 13
  This will be evaluated using the National Adult Reading Test. Participants will be asked to read form a list of 50 words and they will be scored based on whether or not they pronounce each word correctly.

CONTACTS AND LOCATIONS:
Locations (1):
- The Queen Elizabeth Hospital NHS Foundation Trust, Kings Lynn, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Olanrewaju, O. et al. (2022) 'Reducing sedentary behaviour and cognitive function in older people with Mild Cognitive Impairment: Results of a randomized feasibility study', Aging and Health Research, 2(1), p. 100057. doi: https://doi.org/10.1016/j.ahr.2022.100057.